CLINICAL TRIAL: NCT03784495
Title: Is a Combination of Melatonin and Aminoacids Useful to Sarcopenic Elderly Patients? A Randomized Trial
Brief Title: Melatonin Plus Aminoacids for Sarcopenic Elderly
Acronym: MelAASarc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda di Servizi alla Persona di Pavia (Other)
Responsible Party: Principal Investigator, Mariangela Rondanelli, MD, Associate Professor, Azienda di Servizi alla Persona di Pavia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1215/11122015
Record Dates: First submitted 2018-12-14; First posted 2018-12-24 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (P) (Placebo Comparator): Placebo.
  Interventions: Other: Placebo
- Melatonin (M) (Experimental): 1 mg/day of melatonin.
  Interventions: Drug: Melatonin 1mg
- Essential Aminoacids (eAA) (Experimental): 4 g/day of essential aminoacids
  Interventions: Dietary Supplement: Essential Aminoacids (eAA)
- Essential Aminoacids + Melatonin (eAAM) (Experimental): 4 g/day of essential aminoacids and 1 mg/day of melatonin
  Interventions: Combination Product: Essential Aminoacids + melatonin

INTERVENTIONS:
Drug: Melatonin 1mg — 1 mg/day 30 minutes before sleep
  Arms: Melatonin (M)
Dietary Supplement: Essential Aminoacids (eAA) — 4g/day of Essential Aminoacids during breakfast. Packets of powdered amino acid supplements (42.0% leucine, 14.0% lysine, 10.5% valine, 10.5% isoleucine, 10.5% threonine, 7.0% phenylalanine, and 5.5% other) were provided for the participants to be taken with water or milk, and they were instructed to take the 4-gram supplement once a day every day for 4 weeks.
  Arms: Essential Aminoacids (eAA)
Combination Product: Essential Aminoacids + melatonin — 4g/day of Essential Aminoacids during breakfast + 1 mg/day of Melatonin 30 minutes before sleep. Packets of powdered amino acid supplements (42.0% leucine, 14.0% lysine, 10.5% valine, 10.5% isoleucine, 10.5% threonine, 7.0% phenylalanine, and 5.5% other) were provided for the participants to be taken with water or milk, and they were instructed to take the 4-gram supplement once a day every day for 4 weeks.
  Arms: Essential Aminoacids + Melatonin (eAAM)
Other: Placebo — an isocaloric amount of maltodextrin with the same flavor and appearance as the intervention product
  Arms: Placebo (P)

SUMMARY:
To evaluate the effectiveness of melatonin and essential aminoacid supplementation on body composition, protein metabolism, strength and inflammation. The investigators performed a Randomized controlled parallel groups preliminary trial in 159 elderly sarcopenic people (42/117 men/women) assigned to 4 groups: isocaloric placebo (P, n=44), melatonin (M, 1 mg/daily, n=42,), essential aminoacids (eAA 4 g/daily, n=40) or eAA plus melatonin (eAAM, 4 g eAA and 1 mg melatonin/daily, n= 30). The period of intervention was 4 weeks. Data from body composition (DXA), strength (handgrip test) and biochemical parameters for the assessment of protein metabolism (albumin) and inflammation (PRC) were collected at baseline and after the 4-week intervention

ELIGIBILITY:
Inclusion Criteria:

* Aged > or equal 65 years
* Sarcopenic patients, following the Rosetta Study criteria: Skeletal Muscle Index [SMI] was <7.23 kg/m2 in men and <5.45 kg/m2 in women) and loss of strength, evaluated by dynamometer and defined as <30 kg for men and <20 kg for women, using the average value of the two handgrip measurements of the dominant hand.

Exclusion Criteria:

* acute illnesses
* severe liver dysfunction
* severe heart dysfunction
* severe kidney dysfunction
* severe dementia
* uncontrolled diabetes
* dysthyroidism
* any endocrinopathies
* neoplasia
* patients treated with steroids
* patients entirely unable to walk

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 159 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2015-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Total Fat Mass and Total Free Fat Mass (DXA) | 0, 30 days
  Body composition by dual-energy X-ray absorptiometry (DXA). Body composition was measured by DXA, using a Lunar Prodigy DXA (GE Medical Systems, Waukesha, WI). Free Fat mass and Fat mass of specific body regions were measured in kilograms.
Change in Handgrip Strenght | 0, 30 days
  Handgrip strength assessed using a Jamar dynamometer adhering to the standardized protocol recommended by the American Society of Hand Therapists. A weak handgrip was defined as <30 kg for men and <20 kg for women, based on the average value of the two handgrip measurements of the dominant hand

SECONDARY OUTCOMES:
Height | At baseline (0)
  Height measured in meters
Change in Body Weight | 0, 30 days
  Body Weight measured in kilograms
Change in serum proteins | 0, 30 days
  Serum proteins and albumin were measured by automatic biochemical analyzer. They were reported as g/dl
Change in blood lipids (total cholesterol and triglycerides) | 0, 30 days
  Blood lipids (total cholesterol and triglycerides)were measured by automatic biochemical analyzer. They were reported as mg/dl
Change in High-sensitivity C-reactive protein (CRP) | 0, 30 days
  High-sensitivity C-reactive protein (CRP) was expressed in mg/dl.
Change in erythrocyte sedimentation rate (ESR) | 0, 30 days
  Erythrocyte sedimentation rate (ESR) was expressed in mm/hr.
Change in glycaemia | 0, 30 days
  glycemia was expressed in mg/dl
Change in Mini Nutritional Assessment (MNA) | 0, 30 days
  A mini nutritional assessment (MNA) was performed for all participants. The MNA uses 18 questions regarding simple measurements and a brief questionnaire involving an anthropometric assessment (weight, height and weight loss), a general assessment (lifestyle, medication and mobility), and a dietary assessment (number of meals, food and fluid intake, self-assessment of eating autonomy and self-perception of health and nutrition). Every answer give up to a maximum of 3 points. The sum of all points gives the total MNA. A maximum of 30 points can be achieved. A score of ≥ 24 points describes a well-nourished status. A score of 17 to 23.5 points indicates a risk of malnutrition, while less than 17 points indicates malnutrition.
Change in dietary intake | Measures taken at day 1,2,3 and at day 28,29,30
  A trained dietitian used a calibrated dietetic spring scale to weigh all foods served and returned for 3 consecutive days at the beginning and end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Mariangela Rondanelli, Professor, Study Director — IRCCS Mondino Foundation, Pavia
Locations (1):
- Geriatric physical medicine and rehabilitation division at the Istituto Santa Margherita - Azienda di Servizi alla Persona di Pavia, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No
IPD will be not available for other researchers